CLINICAL TRIAL: NCT00107211
Title: A HER-2/Neu Pulsed DC1 Vaccine for Patients With DCIS
Brief Title: Vaccine Therapy in Treating Patients Who Are Undergoing Surgery for Ductal Carcinoma In Situ of the Breast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000416200; UPCC-08102; UPCC-704447
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Vaccines made from peptides and a person's white blood cells may help the body build an effective immune response to kill tumor cells. Injecting the vaccine directly into a lymph node may cause a stronger immune response and kill more tumor cells. Giving vaccine therapy before surgery may be effective treatment for ductal carcinoma in situ of the breast.

PURPOSE: This phase I trial is studying the side effects and best way to give vaccine therapy in treating patients who are undergoing surgery for ductal carcinoma in situ of the breast.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and safety of neoadjuvant ultrasound-guided intranodal vaccine therapy comprising autologous dendritic cells pulsed with recombinant HER2/neu peptides in patients with ductal carcinoma in situ of the breast.
* Determine the sensitization of CD4+ and CD8+ T cells to HER2/neu in patients treated with this vaccine.
* Determine clinical response in patients treated with this vaccine.

Secondary

* Correlate post-vaccine sensitization of CD4+ and CD8+ T cells to HER2/neu with clinical response in patients treated with this vaccine.

OUTLINE: This is a pilot study.

Patients undergo leukapheresis over 2-3 hours to obtain lymphocytes and monocytes. Monocytes are cultured with sargramostim (GM-CSF), interleukin-4, interferon gamma, and lipopolysaccharides for the production of dendritic cells (DC). DC are then pulsed with recombinant HER2/neu peptides to produce the dendritic cell vaccine. Approximately 2 days after leukapheresis, patients receive the vaccine intranodally (into 2 different lymph nodes) by ultrasound guidance once a week for 4 weeks in the absence of unacceptable toxicity. Patients then undergo a second leukapheresis to obtain T lymphocytes for immunologic analysis. Within 2-3 weeks after completion of vaccine therapy, patients undergo lumpectomy or mastectomy AND sentinel lymph node biopsy.

After completion of study treatment, patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal carcinoma in situ (DCIS) of the breast OR DCIS with microinvasion (< 1 mm) by core biopsy or excisional biopsy
* HER2/neu positive tumor, defined as > 10% of the tumor population expressing HER2/neu by immunohistochemical staining
* No evidence of invasive disease by MRI (performed within the past month)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Over 18

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* No thrombocytopenia (i.e., platelet count < 75,000/mm^3)
* No other coagulopathy

Hepatic

* No hepatitis C positivity
* INR > 1.5
* PTT > 50 sec

Renal

* Not specified

Cardiovascular

* Ejection fraction ≥ 50% by MUGA or echocardiogram
* No major cardiac illness

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No HIV positivity
* No toxicity > grade 1
* No other pre-existing medical illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior ipsilateral breast or axillary radiotherapy

Surgery

* No prior ipsilateral axillary dissection
* No prior complete excisional biopsy for DCIS

Other

* No other prior definitive treatment for DCIS
* No concurrent medications that would preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Czerniecki, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States